CLINICAL TRIAL: NCT02169960
Title: Comprehensive Program for Youth Mental Health
Acronym: EMPATHY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Red Deer Public School District (Other); Addiction & Mental Health Strategic Clinical Network (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: AMH-SCN-02
Record Dates: First submitted 2014-06-09; First posted 2014-06-23 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Depression; Suicide; Anxiety
MeSH Terms: conditions — Depression; Suicide; Anxiety Disorders | interventions — Gene Expression; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Middle School, General (Active Comparator): OVK Resiliency Training Program - Cognitive Behavioral Therapy designed to modify negative thoughts and feelings. This program also includes a social problem-solving component.
  Interventions: Behavioral: Resiliency Training
- High School, General (No Intervention): No intervention - no Resiliency training, no online intervention for high school students who do not score at risk for development of mental health issues
- Middle School, Top 10% (Active Comparator): Smart, Positive, Active, Realistic X-factor thoughts (SPARX), Breaking Free, This Way Up online interventions offered to middle school students who score in the Top 10% of their grade for development of mental health issues. OVK Resiliency Training is also provided.
  Interventions: Behavioral: Smart, Positive, Active, Realistic X-factor thoughts (SPARX); Behavioral: Breaking Free; Behavioral: This Way Up; Behavioral: Resiliency Training
- High School, Top 10% (Active Comparator): Smart, Positive, Active, Realistic X-factor thoughts (SPARX), Breaking Free, This Way Up online interventions offered to middle school students who score in the Top 10% of their grade for development of mental health issues.
  Interventions: Behavioral: Smart, Positive, Active, Realistic X-factor thoughts (SPARX); Behavioral: Breaking Free; Behavioral: This Way Up

INTERVENTIONS:
Behavioral: Smart, Positive, Active, Realistic X-factor thoughts (SPARX) — Cognitive Behavioral Therapy based online intervention for depression
  Arms: High School, Top 10%; Middle School, Top 10%
Behavioral: Breaking Free — Online based intervention for Drug and Alcohol Use
  Arms: High School, Top 10%; Middle School, Top 10%
Behavioral: This Way Up — Cognitive Behavioral Therapy online intervention for Depression and Anxiety
  Arms: High School, Top 10%; Middle School, Top 10%
Behavioral: Resiliency Training — Op Volle Kracht (OVK)
  Arms: Middle School, General; Middle School, Top 10%

SUMMARY:
The majority of addiction and mental health problems seen in adults present first in youth. There is strong evidence that prevention and early identification during childhood can mitigate some of these risks. Students who screen at risk for the development of mental illness will be offered online intervention programs with personal guidance from a trained coach. In addition, lessons revolving around resiliency will be provided to all students.

The objectives of this study are:

* Decreased rates of depression and suicide (as well as rates of suicide attempts)
* Decreased use of alcohol, tobacco, and other drugs, with additional downstream benefits such as reduced rates of fetal alcohol spectrum disorder (FASD) and cancer
* Decreased school drop-out rates Decreased rates of interactions with the justice system
* Decreased costs across a range of ministries (health, education, justice, human services), both for youth as well as their families who have been involved in this program

ELIGIBILITY:
Inclusion Criteria:

* The intervention group will be the top 10% of all students participating in the school screening.

Exclusion Criteria:

* Lack of consent, lack of assent, lack of the ability to read and understand the screening tools or intervention tools

Ages: 11 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 5514 (Actual)
Dates: Start 2014-02; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Decrease from baseline in rates of depression and suicide | 12 months
  This will be based on scores on the Patient Health Questionnaire for Adolescents (PHQ-A) questionnaire

SECONDARY OUTCOMES:
Decreased use of alcohol, tobacco and other drugs | Baseline, 3 months, 6 months, 12 months
  Questionnaire (CRAFFT)
Decreased school drop-out rates | 12 months
  Will be tracking the School identification numbers of the students in order to determine how many drop out prior to graduation. This will be compared with historical data from Red Deer Public Schools.
Decreased rates of interactions with the justice system | 12 months
  Will be linking with a data groups' repository as well as ministries in order to determine rates of interactions with the justice system.

CONTACTS AND LOCATIONS:
Overall Officials: Peter H SIlverstone, M.D., Principal Investigator — Alberta Health Services and University of Alberta; Victoria YM Suen, B.A. (hons), Study Director — Alberta Health services
Locations (1):
- Red Deer Public Schools, Red Deer, Alberta, Canada

REFERENCES:
- [Background] Tak YR, Van Zundert RM, Kuijpers RC, Van Vlokhoven BS, Rensink HF, Engels RC. A randomized controlled trial testing the effectiveness of a universal school-based depression prevention program 'Op Volle Kracht' in the Netherlands. BMC Public Health. 2012 Jan 10;12:21. doi: 10.1186/1471-2458-12-21. PMID 22233510
- [Derived] Silverstone PH, Bercov M, Suen VY, Allen A, Cribben I, Goodrick J, Henry S, Pryce C, Langstraat P, Rittenbach K, Chakraborty S, Engels RC, McCabe C. Initial Findings from a Novel School-Based Program, EMPATHY, Which May Help Reduce Depression and Suicidality in Youth. PLoS One. 2015 May 14;10(5):e0125527. doi: 10.1371/journal.pone.0125527. eCollection 2015. PMID 25974146